CLINICAL TRIAL: NCT04224623
Title: Raising Well at Home
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Envolve, Inc., a wholly owned subsidiary of Centene Corporation (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 201510154
Record Dates: First submitted 2020-01-08; First posted 2020-01-13 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Raising Well at Home — The Raising Well at Home intervention was delivered via 3 core home visits designed to be delivered every 4-6 weeks, with additional support via text or phone over 6 months. The home visits were designed to engage the whole family, build skills, and promote changes in the home environment to support lifestyle behavior change. These essential behaviors focused on reducing sugary beverage intake, promoting appropriate portion sizes, improving fruit and vegetable intake, increasing walking and reducing screen time/sedentary activity.

SUMMARY:
The purpose of this pilot study was to test the feasibility and efficacy of a balanced lifestyle intervention for caregivers and their children with obesity, conducted in partnership with Envolve, Inc., a family of comprehensive health solutions and wholly owned subsidiary of Centene Corporation.

DETAILED DESCRIPTION:
This pilot study employed a pretest-posttest design to assess the feasibility and efficacy of the Raising Well at Home pilot intervention delivered by peer coaches on weight (caregiver/child), behaviors (eating, walking), and the home environment. The Raising Well at Home intervention was delivered via home visits with additional support via text or phone over 6 months, beginning after completion of the baseline assessment. This study was implemented in partnership with the parent Raising Well programs located in three states: Florida, Louisiana, and Missouri. The caregiver and the child's height and weight were measured by trained staff in the home with the same scale and stadiometer at the pre- and post-intervention time points. Measures were completed on a paper survey with the same caregiver pre and post intervention delivery.

ELIGIBILITY:
Inclusion Criteria:

* Caregivers had to be at least 18 years old, live in one of the states offering the Raising Well program, and be the primary caregiver to at least one child 2-17 years old served by an Envolve Medicaid Health Plan with International Classification of Diseases, Ninth Revision (ICD-9) coding for overweight or obesity. Caregivers had to be able to give informed consent. If more than one child within a household was eligible to participate, all children were invited to participate.

Exclusion Criteria:

* Unable to speak English or Spanish

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 195 (Actual)
Dates: Start 2016-07-17 (Actual); Primary Completion 2019-08-17 (Actual); Study Completion 2019-08-17 (Actual)

PRIMARY OUTCOMES:
Change in Weight | 6 months
  Mother and child weight assessed by trained staff

CONTACTS AND LOCATIONS:
Locations (1):
- Debra Haire-Joshu, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Haire-Joshu D, Schwarz C, Jacob R, Kristen P, Johnston S, Quinn K, Tabak R. Raising Well at Home: a pre-post feasibility study of a lifestyle intervention for caregivers and their child with obesity. Pilot Feasibility Stud. 2020 Oct 6;6:149. doi: 10.1186/s40814-020-00692-0. eCollection 2020. PMID 33042569